CLINICAL TRIAL: NCT03289676
Title: Determining the Feasibility and Acceptability of a Combined Storytelling Narrative Communication and HIV-tailored Smoking Cessation Intervention for Women Living With HIV
Brief Title: Storytelling Narrative Communication Intervention for Smoking Cessation in Women Living With HIV
Acronym: WISE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Sun S Kim, Associate Professor, University of Massachusetts, Boston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017147
Record Dates: First submitted 2017-09-15; First posted 2017-09-21 (Actual); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Intervention Model Description: : The proposed study has two phases.
  1. Phase 1. Development of Narrative Video: We will first develop narrative videos in collaboration with community organizations of WLHIV in Boston. The video will be filmed in person at the University of Massachusetts Boston.
  2. Phase 2. A Randomized Controlled Trial (RCT) of a Story Telling Narrative Communication Intervention: We will conduct a two-arm RCT assigning participants at a ratio of 1:1 to either one of the two arms (Experimental: HIV-tailored plus SNC interventions vs. Control: HIV-tailored plus attention-control interventions). Both arms will have eight weekly sessions of a 30-minute HIV-tailored cessation intervention (cognitive behavioral therapy plus nicotine patches). All research-related procedures will be conducted remotely.
Who Masked: Outcomes Assessor
Masking Description: The person who assesses follow-up assessments will be blind to treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Quitting Smoking Video (Experimental): This arm will receive a storytelling narrative intervention by watching a video of women living with HIV taking about their success in quitting smoking.
  Interventions: Combination Product: Storytelling Narrative Intervention
- HIV Infection Video (Active Comparator): This arm will watch an attention-control storytelling narrative intervention by watching a video of women living with HIV taking about their life after the diagnosis of HIV.
  Interventions: Combination Product: Storytelling Narrative Intervention

INTERVENTIONS:
Combination Product: Storytelling Narrative Intervention — In the first phase, three sections of a video, each for 5-7 minutes will be produced by "Star" story tellers who are eloquent and have authentic personal experiences of quitting smoking. Participants who receive 8-weekly 30-minute cessation counseling sessions along with NRT are randomly assigned to watch either the smoking cessation video or attention-control video of women taking about their HIV infection.
  Other Names: Cognitive Behavioral Counseling; Nicotine Replacement Therapy

SUMMARY:
HIV has transformed into a chronic illness due to the advent of effective treatments in the absence of a cure. As a result, the prevalence of non-AIDS defining cancers (NADCs), including lung cancer, has increased three-fold among people living with HIV. NADCs now account for 50% of all cancers among the people. Smoking is one of the major contributing factors to lung cancer and smoking prevalence is substantially higher in this population than the general U.S. population. Smoking prevalence does not differ by gender among people living with HIV. Women of color, particularly African American women represent the majority of women living with HIV (WLHIV) followed by Latinas. WLHIV smoke at a rate almost 3 times higher than that for the general U.S. female population (e.g., 42% vs. 16%). The proposed study has two phases: 1) the development of a storytelling narrative communication (SNC) intervention that will be added to an established HIV-tailored smoking cessation intervention and 2) a two-arm randomized controlled trial (RCT) of the HIV-tailored intervention plus the SNC Intervention compared with the HIV-tailored intervention only. The investigators will develop narrative videos with three to five WLHIV who will be talking about their personal struggles with smoking and success in quitting. Preliminary study revealed that the established HIV-tailored intervention was effective only for short-term (≤ 2 months) abstinence. Many relapsed to smoking between the 2nd and 6th month of quitting. The investigators propose that the SNC intervention will be an effective strategy to sustain their quit efforts for long-term abstinence (≥ 6 months). A total of 60 WLHIV will be recruited and randomly assigned to either the experimental arm (a combination of HIV-tailored and SNC interventions) or the control arm (HIV-tailored intervention only). Specific aims of the study are to 1) Identify SNC intervention components that are rated high in transport and identification for use as an enhancement to an HIV-tailored smoking cessation intervention; 2) Determine the feasibility and acceptability of the SNC intervention for WLHIV by assessing the rate of recruitment and retention for feasibility and the degree of transport and identification for acceptability; and 3) Establish an effect size of HIV-tailored and SNC interventions for smoking cessation in comparison with the HIV-tailored smoking cessation intervention only for WLHIV, for subsequent grant applications.

DETAILED DESCRIPTION:
The proposed study employs a mixed-methods research design. The investigators will first develop narrative videos in collaboration with community organizations of WLHIV in Boston. Second, the investigators will conduct a two-arm RCT assigning participants at a ratio of 1:1 to either one of the two arms (Experimental: HIV-tailored plus SNC interventions vs. Control: HIV-tailored intervention). Both arms have eight weekly sessions of a 30-minute HIV-tailored cessation intervention (cognitive behavioral therapy plus nicotine patches). The experimental arm will receive three 5-7 minute SNC videos, each per month between the first and third month of quitting, whereas the control arm will receive three 5-minute attention control videos at the same monthly interval.

A total of 60 WLHIV will be recruited via online and offline advertisements and personal networks of community organizations and health care providers who work for people with HIV. To participate in the study, the following criteria must be met: women who 1) are able to speak English; 2) self-report HIV infection and submit a supplementary document if necessary; 3) are between the ages of 18 and 65; 4) have been smoking at least 5 cigarettes a day for the past 6 months; 5) own a mobile phone with an access to a video call application such as Skype, Imo, Tango, and Face Time; 6) are willing to quit smoking within the next 4 weeks from the baseline assessment; and 7) agree to use an approved form of birth control (e.g., oral medications, condoms, and intrauterine devices) during the study period. Individuals will be excluded if they: 1) are not able to speak English; 2) are pregnant or lactating; 3) have an active skin disease or serious alcohol use problems (≥ 26 on the Alcohol Use Disorders Identification Test), 4) self-report currently receiving treatment for a serious mental illness (e.g., schizophrenia and bipolar disorder); or 5) currently use any illegal substances excluding marijuana.

The investigators will recruit participants with frequent announcements of the study in Craigslist and paid online advertisements. The majority of intake interviews will be conducted via telephone, which will take 30 minutes at most. To prevent attrition, the investigators will execute several strategies, including tracking subjects at least every other month and providing incentives for follow-up testing. Counselors will proactively call participants prior to each therapy session and confirm the appointment a few hours before the session. A research assistant (RA) who will be blinded to the intervention condition will conduct all follow-up assessments via telephone calls and videoconferencing for saliva cotinine tests.

ELIGIBILITY:
Inclusion Criteria:

women who:

1. are able to speak English
2. self-report HIV infection and submit a supplementary document if necessary
3. are between the ages of 18 and 65
4. have been smoking at least 5 cigarettes a day for the past 6 months
5. own a mobile phone with an access to a video call application such as Skype, Imo, Tango, and Face Time
6. are willing to quit smoking within the next 4 weeks from the baseline assessment; and
7. agree to use an approved form of birth control (e.g., oral medications, condoms, and intrauterine devices) during the study period.

Exclusion Criteria:

Women who:

1. are not able to speak English
2. are pregnant or lactating
3. have an active skin disease or serious alcohol use problems (≥ 26 on the Alcohol Use Disorders Identification Test59)
4. self-report currently receiving treatment for a serious mental illness (e.g., schizophrenia and bipolar disorder) or
5. currently use any illegal substances excluding marijuana.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Who are biologically females.
Enrollment: 53 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun S Kim, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University Massachusetts Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim SS, DeMarco RF. The Intersectionality of HIV-Related Stigma and Tobacco Smoking Stigma With Depressive and Anxiety Symptoms Among Women Living With HIV in the United States: A Cross-sectional Study. J Assoc Nurses AIDS Care. 2022 Sep-Oct 01;33(5):523-533. doi: 10.1097/JNC.0000000000000323. Epub 2022 Jan 7. PMID 34999667
- [Derived] Kim SS, Cooley ME, Lee SA, DeMarco RF. Prediction of Smoking Abstinence in Women Living With Human Immunodeficiency Virus Infection. Nurs Res. 2020 May/Jun;69(3):167-175. doi: 10.1097/NNR.0000000000000421. PMID 31977840
- [Derived] Kim SS, Lee SA, Mejia J, Cooley ME, Demarco RF. Pilot Randomized Controlled Trial of a Digital Storytelling Intervention for Smoking Cessation in Women Living With HIV. Ann Behav Med. 2020 May 25;54(6):447-454. doi: 10.1093/abm/kaz062. PMID 31863582

RESULTS

PARTICIPANT FLOW:
Groups:
- Quitting Smoking Film: This arm viewed a storytelling narrative film of six women living with HIV taking about their success in quitting smoking.
  A total of 27 women were randomized into this arm and four women withdrew from the study right before receiving any of the allotted intervention.
  Of the remaining 23 women, 18 women received at least 80% of the allotted intervention, and all 23 women completed the study without any more loss.
  Outcome analysis was done separately with 27 women who were randomized into the arm and with 23 women who actually received any part of the allotted intervention.
- HIV Infection (an Attnetion-control) Film: This arm will watch an attention-control storytelling narrative intervention by watching a video of women living with HIV taking about their life after the diagnosis of HIV.
  A total of 26 women were randomized into this arm and 20 women received at least 80% of the allotted intervention. One was lost during the follow-up period and 25 women completed the study.
  Outcome analysis was done with 26 women who were randomized into the arm.
Period: Overall Study
Arm/Group | Quitting Smoking Film | HIV Infection (an Attnetion-control) Film
Started | 27 | 26
Completed (Received 80% of the allotted intervention) | 23 | 25 (Received 80% of the allotted intervention)
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Quitting Smoking Video: This arm watched a film in which six women living with HIV talk about why they decided to quit smoking and how they did.
- HIV Infection Video: This arm watched an attention-control film in which four women talk about their everyday lives before and after the diagnosis of HIV.
- Total: Total of all reporting groups
Arm/Group | Quitting Smoking Video | HIV Infection Video | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.81 (7.02) | 50.92 (6.76) | 51.38 (6.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 53
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 24 | 46
  White | 1 | 2 | 3
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 1
Fagerstrom Test for Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — The scale has 6 items with four dichotomous items and two 4-point items. Its total score is the sum of each item score and ranges 0 to 10. The higher values represent a worse outcome.
  units on a scale | 6.19 (2.42) | 4.73 (2.16) | 5.47 (2.39)

OUTCOME MEASURES:

1. Primary Outcome: Adherence Rate
Description: Women in both arms who reported having watched all four videos of the storytelling narrative intervention.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Quitting Smoking Video | HIV Infection Video
Number analyzed (Participants) | 23 | 25
Participants | 20 | 17
Statistical Analysis 1: Comparison: Quitting Smoking Video vs HIV Infection Video; Test type: Superiority; p = 0.29, Fisher Exact

2. Primary Outcome: 3-month Abstinence Rate
Description: Participants in both arms who self-reported having not smoked a cigarette for 3 months from the quit day and also whose salivary cotinine test showed a negative result at 3-month follow-up.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Quitting Smoking Video | HIV Infection Video
Number analyzed (Participants) | 27 | 26
Participants | 10 | 4

3. Secondary Outcome: Self-efficacy in Resisting Smoking Temptation.
Description: This scale assesses participants' confidence (self-efficacy) in resisting smoking temptation in nine specific situations. Each item score ranges from 1 (completely unconfident) to 5 (completely confident). The scale score is the sum of each item score and ranges from 9 to 45. Higher scores represent more confidence and better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on the scale
Arm/Group | Quitting Smoking Video | HIV Infection Video
Number analyzed (Participants) | 23 | 25
units on the scale | 35.5 (10.1) | 31.8 (8.1)
Statistical Analysis 1: Comparison: Quitting Smoking Video vs HIV Infection Video; Test type: Other; p = 0.029, Regression, Logistic; Odds Ratio, log = 1.12, 95% CI 2-sided [1.00 to 1.24]

ADVERSE EVENTS:
Time Frame: 4 months
Groups:
- Quitting Smoking Video: This arm received a storytelling narrative intervention by watching a video of women living with HIV taking about their success in quitting smoking.
- HIV Infection Video: This arm watched an attention-control storytelling narrative intervention by watching a video of women living with HIV taking about their life after the diagnosis of HIV.
Arm/Group | Quitting Smoking Video | HIV Infection Video
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 0/27 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT03289676/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT03289676/SAP_001.pdf
  • Informed Consent Form (2018-02-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT03289676/ICF_002.pdf